CLINICAL TRIAL: NCT00418912
Title: Family Study in Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Raz Gross, Head, Mental Health Epidemiology, The Gertner Institute for Epidemiology
Other Study IDs: SHEBA-06-4329-RG-CTIL
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Schizophrenia; Family; Genetics
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective

SUMMARY:
Schizophrenia is a severe mental illness which is considered to have, among other, a genetic etiology. One of the most efficient tools in genetic-psychiatry is the investigation of multiplex families.

The current study will identify patients of multiplex families and to map their family connections and the presence of mental illnesses among family members.

ELIGIBILITY:
Inclusion Criteria:

1. Schizophrenia
2. Multiplex family
3. Able to understand and sign the informed concent form.
4. Hebrew speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-12 (Estimated); Study Completion 2009-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Raz Gross, MD, Principal Investigator — Mental Health Epidemiology & Psychosocial Aspects of Illness, The Gertner Institute for Epidemiology and Health Policy Research, Sheba Medical Center, Tel Hashomer , Israel; Michael Bunzel, MD, Study Director — Psychiatric Unit, Sheba Medical Center, Tel Hashomer, Israel
Locations (2):
- Israel (2):
  - Psychiatric unit, Sheba Medical Center, Tel Litwinsky
  - Seba Medical Center, Tel Litwinsky